CLINICAL TRIAL: NCT05124288
Title: Analysis of the Immunobiology of Acute Myeloid Leukemia Relapses After Hematopoietic Stem Cell Transplant (HSCT) for the Generation of Guidelines and Personalized Therapeutic Pathways
Brief Title: Analysis of the Immunobiology of Acute Myeloid Leukemia Relapses After Allogeneic Hematopoietic Stem Cell Transplant (HSCT) for the Generation of Guidelines and Personalized Therapeutic Pathways
Acronym: GITMO-RELAPSE
Status: Recruiting | Type: Observational
Sponsor: Ciceri Fabio (Other)
Collaborators: Gruppo Italiano Trapianto di Midollo Osseo (Other); Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor-Investigator, Ciceri Fabio, Principal Investigator, Professor and Head of Hematology, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: GITMO-RELAPSE
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia, in Relapse
Keywords: Haematopoietic Stem Cell Transplantation; Graft versus Host Disease; Acute Myeloid Leukemia; Human Leukocyte Antigens loss
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral and bone marrow blood, withdrawn during clinical practice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute Myeloid Leukemia relapsed patients: Adult patients (< 18 years old), with Acute Myeloid Leukemia, who relapse after allogeneic transplantation from either family or unrelated donors, regardless of the cellular source of the transplant (bone marrow, mobilized peripheral stem cells or cord blood).
  Interventions: Other: Observations on Relapsed AML Allogeneic Transplanted patients

INTERVENTIONS:
Other: Observations on Relapsed AML Allogeneic Transplanted patients — This is not an interventional clinical study. This is a retrospective/prospective observational study on Relapsed AML Allogenic Transplanted patients. Additional samples will be collected during the standard practice.

SUMMARY:
This is a retrospective and prospective non-interventional multicenter observational study. Neither diagnostic approaches nor experimental drugs/procedure will be applied and the samples will take place at the same time as the samples will be taken during routinary clinical practice.

The aim of this study is to analyze the immunobiology of Acute Myeloid Leukemia (AML) relapses after allogeneic HSCT for the generation of guidelines and personalized therapeutic pathways.

DETAILED DESCRIPTION:
Background: The identification of leukemic relapses characterized by the "Human Leukocyte Antigens loss" event or by changes in the expression levels of genes involved in antigen presentation and lymphocyte co-stimulation demonstrate how a complete characterization of disease recurrence is necessary to ensure the patient a treatment that is as personalized and targeted as possible, avoiding the choice of sub-optimal or, sometimes, harmful therapies. Unfortunately, the identification of the post-transplant relapse mechanism is now far from being part of an established clinical routine, mainly due to the lack of quick and easy-to-access diagnostic tools and multicentre studies demonstrating the efficacy of a type of personalized therapeutic approach.

The main objective of the study is to favor, exploiting the consolidated collaboration between the Italian transplant centers belonging to the Italian Group of Bone Marrow Transplantation, Hematopoietic Stem Cells and Cell Therapies (GITMO), the implementation in clinical practice of an in-depth biological study of relapses of leukemia in order to allow an increasingly targeted and effective planning of the therapeutic strategies to be implemented, ensuring better patient survival.

The study is divided into two parts:

* data collection, from clinical standard practice, of patients with relapse of the disease which will allow to standardize the therapeutic management process and will allow us to promote innovative clinical studies on acute myeloid leukemia post allogeneic HSCT, with the ultimate aim of improving the survival of these patients;
* biological substudy that will allow to define the role of the tumor microenvironment in promoting or counteracting the phenomenon of relapse by identifying its specific alterations in the various forms of disease relapse.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Acute Myeloid Leukemia, who relapse after allogeneic transplantation from either family or unrelated donors, regardless of the cellular source of the transplant (bone marrow, mobilized peripheral stem cells or cord blood), who have signed the informed consent of the study;
* For the coordinating center, all patients who have previously signed informed consent to the "Hematological Neoplasms Biobank" and for which samples, stored in the Biobank are available.
* For the other centers, all patients who have previously signed an informed consent, aimed at the prior authorization for the storage of samples in the biobank of the aforementioned center, according to centers own practice, and for which samples, stored in a Biobank, are available.

Exclusion Criteria:

* Participation in clinical protocols that expressly exclude the possibility of participating in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort of this study will be composed of adult patients with Acute Myeloid Leukemia, who will relapse after allogeneic transplantation from either familial or unrelated donor, regardless of the cellular source of the transplant (bone marrow, mobilized peripheral stem cells or cord blood).
  The samples of interest are those taken at the time of post-transplant recurrence at the same time as routine investigations and may be of both medullary blood and peripheral blood, as long as the samples have a percentage of pathological cells equal to at least 5% of cellularity.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | From date of transplant infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  The probability of disease-free survival will be calculated from the transplant infusion time to the date of death, last follow-up and / or disease recurrence / progression.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Yet to be determined